CLINICAL TRIAL: NCT02367703
Title: Assessment of Feasibility and Benefit of the Use of Less Than 3 Millimeter Diameter's Instruments Compared to Standard Size Instruments in Laparoscopic Hysterectomy: a Randomized Single-center Comparative Study
Brief Title: Feasibility and Benefit of Laparoscopic Hysterectomy With Less Than 3 Millimeter Diameter's Instruments in Current Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: STORZ® laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0223; 2014-A01698-39 (Other: ANSM)
Record Dates: First submitted 2015-02-06; First posted 2015-02-20 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Benign Uterine Diseases
Keywords: Mini-laparoscopy; hysterectomy; Benign uterine diseases; Operative time

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- standard instrument (Experimental): That is why we propose a randomized comparative study between standard instrument and less than 3 millimeter diameter's instruments to achieve in daily practice laparoscopic hysterectomy
  Interventions: Procedure: laparoscopic hysterectomy
- less than 3 millimeter diameter's instruments (Other): That is why we propose a randomized comparative study between standard instrument and less than 3 millimeter diameter's instruments to achieve in daily practice laparoscopic hysterectomy
  Interventions: Procedure: laparoscopic hysterectomy

INTERVENTIONS:
Procedure: laparoscopic hysterectomy

SUMMARY:
Hysterectomy for benign uterine disease is often intended to young perimenopausal patients. Currently laparoscopic hysterectomy is commonly used in this indication. We are wondering if decreasing the diameter of laparoscopic instruments could reduce postoperative pain and improve esthetic result without increasing operative time. The purpose of the study is to improve patients' care.

DETAILED DESCRIPTION:
That is why we propose a randomized comparative study between standard instrument and less than 3 millimeter diameter's instruments to achieve in daily practice laparoscopic hysterectomy.

The study will be unicentric, single-blind. Study period will be one year and 4 months. Patients will be enrolled in pre-operative consultations or at the weekly staff. They will have to sign an informed consent.

The day before surgery: patients will be randomized by the statistician. A resident will carry out a preoperative ultrasound to determine an estimated uterine volume. Nurses will make a blood test (hemoglobin).

The day of surgery we will assess: operative time, surgeon's ergonomics, the amount of bleeding, patient's pain at rest and mobilization.

At Day-1 post surgery nurses will make an other blood test (hemoglobin) and we will assess patient's pain at rest and mobilization.

At the postoperative consultation we will lister : complications (Accordion Severity score classification), esthetic result (PSAQ), patient's pain.

ELIGIBILITY:
Inclusion Criteria:

* patient candidate for total inter-adnexal hysterectomy or for hysterectomy with oophorectomy and
* benign gynecological pathology: fibroids, adenomyosis, polyps, dysfunctional uterine bleeding.

and

* affiliation to social security and
* informed consent

Exclusion Criteria:

* ASA III or IV patients,
* age> 80 years old,
* history of major abdominal surgery by laparotomy
* severe obesity (BMI> 35kg / m2)
* pathology of hemostasis and coagulation (liver disease, bleeding disorders)
* uterine volume estimated on preoperative ultrasonography > 300 g
* minor patients,
* adult lacking legal capacity
* patients suffering from mental illness incompatible with informed consent, refusal to participate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
operative time | at day 1 (at the end of the surgery)

SECONDARY OUTCOMES:
quantity of intraoperative bleeding | at day 1 (at the end of the intervention)
hemoglobin | at day 1
Pain Rating Scale (VAS) | at day 1 (at 6 hours potoperative hours)
Pain Rating Scale (VAS) | at day 1 (at 24 postoperative hours)
standard laparoscopy conversion rate | at day 1
postoperative complications | at each additional hospitalisation
  postoperative complications according Accordion Severity Classification score (grade> or = 2) listed at each additional hospitalisation
Patient Scar Assessment Scale (PSAS) | at 6 and 8 weeks after surgery.
  Patient Scar Assessment Scale (PSAS)completed at the time of post-operative consultation
Surgen's ergonomics | at the end of the surgery
  Surgen's ergonomics evaluated at the end of the surgery (NASA-TLX scale)

CONTACTS AND LOCATIONS:
Overall Officials: Revaz BOTCHORISHVILI, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France